CLINICAL TRIAL: NCT07323147
Title: Clinical Efficacy of Exoskeleton Robot-Assisted Rehabilitation on Lower Limb Functional Recovery in Elderly Patients With Hip Fracture: A Multicenter, Open-Label, Randomized Controlled Clinical Trial
Brief Title: Clinical Efficacy of Exoskeleton Robot-Assisted Rehabilitation on Lower Limb Functional Recovery in Elderly Patients With Hip Fracture
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hai bao (Other)
Responsible Party: Sponsor-Investigator, Hai bao, Attending Physician, Beijing Jishuitan Hospital
Organization: Beijing Jishuitan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: JST-IIT-2025086
Record Dates: First submitted 2025-12-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hip Fracture; Geriatrics; Lower Extremity Dysfunction; Postoperative Rehabilitation; Gait Disorders
Keywords: Exoskeleton Robot; Robotic Rehabilitation; Wearable Devices; Randomized Controlled Trial; Multicenter Study; Recovery of Function; Harris Hip Score
MeSH Terms: conditions — Hip Fractures; Mobility Limitation | interventions — Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: The target total sample size is 86 participants. A competitive enrollment model will be used, with no pre-set quota for individual study sites. All participating centers will collectively compete to achieve the overall recruitment target.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Training with exoskeleton+Conventional rehabilitation program
  Interventions: Device: Exoskeleton
- Control Group (Active Comparator): Conventional rehabilitation program
  Interventions: Other: Conventional rehabilitation program

INTERVENTIONS:
Device: Exoskeleton — 1. Postural Adaptation Training: With exoskeleton support, the patient transitions from a lying or sitting position to an upright stance and maintains this posture for a prescribed duration.
  2. Range of Motion (ROM) and Flexibility Training: The robot guides the patient's lower limbs (hip, knee, and ankle joints) through passive, large-amplitude flexion and extension movements within a safe range.
  3. Muscle Reactivation and Low-Intensity Strengthening: With robotic assistance, the patient actively attempts to execute joint flexion and extension movements. The exoskeleton provides adjustable assistance levels proportionate to the patient's muscular capacity.
  Arms: Intervention Group
Other: Conventional rehabilitation program — 1. Based on the patient's general condition and baseline status, ankle pumps, and isometric contractions of the quadriceps and gluteus medius will be performed progressively according to current international and domestic rehabilitation guidelines; followed by initiation of knee extension exercises, hip abduction exercises of the affected limb, and bridge exercises;
  2. Once the patient's physical capacity has recovered to a relatively stable level, progressive resistance training for the quadriceps, hamstrings, and gluteal muscles will be gradually introduced, along with concurrent strength training for both upper limbs and the unaffected lower limb;
  3. Depending on the patient's rehabilitation progress, training in position transfer, standing, and gait will be initiated; traditional physical rehabilitation modalities such as therapeutic cycling, electrical stimulation, and medium-frequency therapy devices may also be incorporated.
  Arms: Control Group

SUMMARY:
With the intensification of population aging, hip fracture, as a common bone disease, is seeing an increasing incidence rate among the elderly population. Traditional rehabilitation training methods can no longer fully meet the functional recovery needs of elderly patients with hip fractures. Due to their wearability and intelligence, exoskeleton robots provide an innovative solution for rehabilitation training. This study aims to explore the application effects of exoskeleton robots in postoperative rehabilitation for elderly patients with hip fractures by utilizing exoskeleton robot-assisted rehabilitation training for elderly hip surgery patients. The focus is on its improvements in motor ability, balance ability, and pain levels, while also assessing its impact on patients' overall quality of life and the prevention of complications.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or older, regardless of gender.
* Diagnosed with a unilateral hip fracture resulting from low-energy trauma by imaging (X-ray/CT), and having undergone surgical treatment (internal fixation or arthroplasty).
* The participant or their legal guardian understands and agrees to participate in the clinical trial and is willing to provide voluntary written informed consent.

Exclusion Criteria:

* Life expectancy of less than 6 months.
* History of neurological disorders such as prior stroke, spinal cord injury, Parkinson's disease, or myasthenia gravis.
* Severe joint contractures, deformities, or heterotopic ossification in the lower limbs that would prevent proper device fitting.
* Body weight exceeding the device's maximum load capacity (>100 kg).
* Height outside the adjustable range of the device.
* Presence of a pathological fracture or multiple fragility fractures.
* Presence of severe osteoarthritis or trauma in the contralateral lower limb that significantly impairs function.
* Comorbidities including active malignancy or systemic infection.
* Comorbidities such as thromboembolic disease in the lower limbs, pneumonia, or pressure injuries (bedsores).
* Comorbidities affecting rehabilitation capacity, including unstable angina, heart failure, severe sequelae of stroke, severe chronic obstructive pulmonary disease (COPD), or severe hepatic/renal dysfunction.
* Poor compliance, cognitive impairment preventing cooperation, or diagnosed psychiatric disorders such as depression or anxiety.
* Participation in any other clinical trial within the 3 months prior to screening.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 1-month post-intervention (T1), 3-month post-intervention (T2).
  Assessed using the Harris Hip Score (HHS), a disease-specific instrument widely used for evaluating outcomes following hip surgery or in hip pathology. The scale assesses the patient across four domains: pain (44 points), function (47 points), range of motion (5 points), and absence of deformity (4 points). The total score ranges from 0 to 100 points. A higher score indicates better hip joint function and less disability. The reported value is the total HHS score (points).

SECONDARY OUTCOMES:
Berg Balance Scale | 1-month post-intervention (T1), 3-month post-intervention (T2)
  Assessed using the Berg Balance Scale. This scale consists of 14 items that evaluate static and dynamic balance abilities (e.g., standing, turning, picking up objects). Each item is scored from 0 to 4 points. The total score ranges from 0 to 56 points. A higher score indicates better balance function. The reported value is the total scale score (points).
Timed Up and Go Test | 1-month post-intervention (T1), 3-month post-intervention (T2).
  The time required for the subject to rise from a chair, walk 3 meters, turn around, walk back, and sit down is recorded. The reported value is the time to complete the test (seconds). A shorter time indicates better functional mobility.
6-Minute Walk Test | 1-month post-intervention (T1), 3-month post-intervention (T2).
  The maximum distance a subject can walk on a flat surface within 6 minutes is measured. The reported value is the total walking distance (meters). A greater distance indicates better walking endurance.
Visual Analogue Scale (VAS) | 1-month post-intervention (T1), 3-month post-intervention (T2).
  Assessed using the Visual Analogue Scale (VAS) to evaluate the subject's average pain intensity over the past 24 hours. Subjects mark their pain level on a 10-cm line anchored with "no pain" (0) and "worst pain imaginable" (10). The reported value is the distance from the start point to the mark (centimeters). A higher score indicates more severe pain.
Range of Motion Measurement | 1-month post-intervention (T1), 3-month post-intervention (T2).
  The active range of flexion of the affected hip joint is measured using a universal goniometer. The reported value is the angle of flexion (degrees). A greater angle indicates better joint mobility function.
Psychological Assessment | Baseline (T0), 1-month post-intervention (T1), 3-month post-intervention (T2).
  Assessed using the anxiety subscale (HADS-A) of the Hospital Anxiety and Depression Scale (HADS). This subscale comprises 7 items, each scored from 0 to 3 points. The total score ranges from 0 to 21 points. A higher score indicates more severe anxiety symptoms. The reported value is the total subscale score for anxiety (points).
Proteomics Analysis | Baseline (T0), 1-month post-intervention (T1), 3-month post-intervention (T2).
  Proteomic analysis is performed on fasting venous blood samples to compare protein expression profiles between different time points (T1/T2 vs. T0) and between groups (intervention vs. control). The reported value is the number of statistically significant differentially expressed proteins identified under set significance thresholds (e.g., p<0.05 and fold change >1.5).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Jishuitan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be publicly shared due to ethical and privacy considerations, institutional data use agreements, and current resource limitations. Access may be reconsidered in compliance with future funder or publisher requirements. For inquiries, please contact the principal investigator.